CLINICAL TRIAL: NCT04523896
Title: High-Dose-Rate Prostate Brachytherapy Combined With Stereotactic Ablative Prostate Radiotherapy for Patients Diagnosed With Intermediate and High-risk Prostate Cancer. Phase II Clinical Trial.
Brief Title: HDR Brachytherapy Plus Stereotactic Ablative Prostate Radiotherapy for Patients With Intermediate and High-risk Prostate Cancer
Acronym: BRAchySABR
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: David Büchser (Other Government)
Responsible Party: Sponsor-Investigator, David Büchser, Radiation Oncology Consultant, Principal Investigator., Biobizkaia Health Research Institute
Organization: Biobizkaia Health Research Institute (Other Government)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BRAchySABR
Record Dates: First submitted 2020-08-11; First posted 2020-08-24 (Actual); Last update posted 2020-08-24 (Actual); Status verified 2020-08

CONDITIONS: Prostatic Neoplasm
Keywords: High-Dose-Rate brachytherapy; SABR; SBRT; Quality of life
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: Single Group Assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HDR brachytherapy + SABR (Experimental): High-Dose-Rate prostate brachytherapy: a single fraction of 15 Gy to the whole prostate.
  Between 2-4 weeks after the brachytherapy session, SABR treatment will be delivered:
  5 sessions of 5 Gy in consecutive days (i.e monday to friday) to a total dose of 25 Gy to the whole prostate.
  Interventions: Radiation: Real time High-Dose-Rate prostate brachytherapy in combination with stereotactic prostate radiotherapy

INTERVENTIONS:
Radiation: Real time High-Dose-Rate prostate brachytherapy in combination with stereotactic prostate radiotherapy — - Brachytherapy: Real time HDR prostate brachytherapy using a MRI-trans-rectal ultrasound image fusion protocol: single fraction of 15 Gy.
  Planning software: Oncentra prostate (Nucletron)
  - External beam radiotherapy: Stereotactic ablative radiation therapy (SABR): 5 session in 5 consecutive days, 5 Gy per fraction to the prostate.
  Intra-fraction gold seeds monitoring using Auto beam Hold solution (Varian) Planning software: Eclipse (Varian).
  Other Names: HDR brachytherapy; SABR; SBRT

SUMMARY:
Dose escalation is nowadays a standard strategy in radiotherapy for prostate cancer. Besides, it is believed that due to the radiobiology characteristics of prostate cells (low alpha/beta ratio), the delivery of higher radiation doses per fraction could theoretically improve the efficacy of the treatment. In this context, the combination of prostate brachytherapy and external beam radiotherapy (EBRT) has proven to be the most effective method of dose escalation significantly improving disease control in randomized clinical trials. Unfortunately, this strategy is also associated with an increased risk of acute and late adverse events compared to conventional EBRT alone. It has been proposed that this increase in adverse events could be related to the use Low-Dose-Rate (LDR) brachytherapy and that High-Dose-Rate (HDR) brachytherapy (a more modern and accurate procedure) could reduce this risk.

On the other hand, Stereotactic Ablative Radiotherapy (SABR) is a high-precision radiation technique that allows the delivery of higher doses per fraction in fewer sessions, reducing the total treatment time.

The investigators hypothesized that the combination of two highly conformal radiation techniques (HDR brachytherapy and SABR) could be well tolerated, while reducing total treatment time and therefore improving patient quality of life.

This is a single arm Phase II clinical trial designed to test the feasibility, tolerability and impact on quality of life of the combination of High-Dose-Rate prostate brachytherapy and SABR for patients with intermediate and high-risk prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of adenocarcinoma of the prostate.
* Intermediate or high-risk disease (as per NCCN criteria):

  * Intermediate risk:
* Clinical stage ≤ T2c
* Gleason score 7 and initial PSA ≤ 20 ng/ml.
* Gleason score ≤ 6 and initial PSA > 10 and ≤ 20 ng/ml.

  * High risk,at least one of the following:
* Clinical stage T3a-b.
* Gleason score 8-10.
* Initial PSA > 20 ng/ml.
* Life expectancy of more than 10 years
* Able and willing to complete Expanded Prostate Index Composite (EPIC) end EORTC questionnaires
* Eastern Cooperative Oncology Group (ECOG) of 0 - 2.
* Willing to give informed consent to participate in this clinical trial
* Give competent informed consent to participate in this trial.

Exclusion Criteria:

* Documented nodal or distant metastases.
* Previous pelvic radiotherapy.
* Clinical stage T4.
* Clinical stage T3a or T3b in which the coverture of the extraprostatic disease is not feasible (as deemed by the treating physician).
* Prostate volume > 70 cc (measured on MRI).
* Poor baseline urinary function defined as International Prostate Symptom Score (IPSS) >17
* Contra-indication to radical prostate radiotherapy
* Significant medical co-morbidity rendering patient unsuitable for general anaesthetic

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-07-01 (Actual); Primary Completion 2021-07 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
Deterioration of patient quality of life as assessed by EPIC-26 (The Expanded Prostate Cancer Index Composite short form) | 24 months
  Impact on Quality of life affecting the genitourinary, gastrointestinal, sexual and hormonal domains using the EPIC-26 short form (graded from 0-100, with higher scores representing better quality of life). Baseline value (i.e. prior to treatment) will be compared to values recorded 1 month, 3 months, 12 months and 24 months after treatment.
Deterioration of patient quality of life as assessed by EORTC (European Organisation for Research and Treatment of Cancer) QLQ-PR25 short form. | 24 months
  Impact on Quality of life affecting the genitourinary, gastrointestinal, sexual and hormonal domains using the EORTC QLQ-PR25 short form (items and scale scores of the QLQ-PR25 are linearly transformed to a 0-100 scale, with higher scores reflecting either more symptoms (urinary, bowel, hormonal treatment-related symptoms) or higher levels of functioning (sexual).). Baseline value (i.e. prior to treatment) will be compared to values recorded 1 month, 3 months, 12 months and 24 months after treatment.
Incidence and severity of genitourinary treatment-related acute adverse events graded according to CTCAE (Common Terminology Criteria for Adverse Events) v5.0 scale. | 3 months
  Every urinary event occurring within 3 months from treatment completion will be defined as "acute event". All adverse events will be recorded and graded according to CTCA V5.0 scale (graded from 0-5 with greater values representing worse outcomes)
Incidence and severity of gastrointestinal treatment-related acute adverse events graded according to CTCAE (Common Terminology Criteria for Adverse Events) v5.0 scale. | 3 months
  Every gastrointestinal event occurring within 3 months from treatment completion will be defined as "acute event". All adverse events will be recorded and graded according to CTCA V5.0 scale (graded from 0-5 with greater values representing worse outcomes)
Incidence and severity of genitourinary treatment-related late adverse events graded according to CTCAE (Common Terminology Criteria for Adverse Events) v5.0 scale. | 24 months months
  Every genitourinary event occurring 3 months after treatment completion will be defined as "late event". All adverse events will be recorded and graded according to CTCA V5.0 scale (graded from 0-5 with greater values representing worse outcomes) 6 months, 12 months and 24 months after treatment.
Incidence and severity of gastrointestinal treatment-related late adverse events graded according to CTCAE (Common Terminology Criteria for Adverse Events) v5.0 scale. | 24 months months
  Every gastro-intestinal event occurring 3 months after treatment completion will be defined as "late event". All adverse events will be recorded and graded according to CTCA V5.0 scale (graded from 0-5 with greater values representing worse outcomes) 6 months, 12 months and 24 months after treatment.

SECONDARY OUTCOMES:
Treatment efficacy in biochemical control measured through PSA (prostate specific antigen) level. | 24 months
  PSA will be evaluated at baseline and in every follow-up visit (1 month, 3 months, 6 months, 12 months and 24 months after treatment completion.

CONTACTS AND LOCATIONS:
Overall Officials: David Büchser, MD, Principal Investigator — Biocruces Bizkaia Health Research Institute/ Cruces University Hospital; Alfonso Gomez-Iturriaga, MD, PhD, Principal Investigator — Biocruces Bizkaia Health Research Institute/ Cruces University Hospital
Locations (1):
- Biocruces Bizkaia Health Research Institute/Cruces University Hospital, Barakaldo, Bizkaia, Spain

IPD SHARING:
Plan to Share IPD: No